CLINICAL TRIAL: NCT06060873
Title: Phase II Trial of Serum Micro RNA-371 in Detecting Active Germ Cell Tumors in Patients With Suspected Regional Disease - (MAGESTIC Trial: MiRNA in Detecting Active Germ Cell Tumors in Early Suspected and MetastaTIC Disease Trial)
Brief Title: MAGESTIC Trial: MiRNA in Detecting Active Germ Cell Tumors in Early Suspected and MetastaTIC Disease Trial
Status: Suspended | Type: Observational
Why Stopped: Asking FDA for risk determination status
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4T-22-2; NCI-2023-00412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4T-22-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Malignant Testicular Germ Cell Tumor
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: This cohort involves all CS-I GCT patients which is defined as GCT in orchiectomy specimen (seminoma and NSGCT), normal conventional staging imaging, and normal/low stable tumor markers. The current standard of care for management of CS-I disease is either surveillance, RPLND, or systemic therapy. Surveillance is preferred however is largely dependent on clinician discretion. In this cohort miRNA-371 level will be drawn at any timepoint after orchiectomy. Patient will continue to be followed with miRNA levels with each conventional marker draw until 2 years, and followed according to standard of care guidelines until 5 years.
  Interventions: Other: Clinical Stage I Disease
- Cohort 2: This cohort involves all GCT patients with radiographically enlarged retroperitoneal lymph nodes <3 cm (initial CS-I GCT patients with radiographic evidence of retroperitoneal lymph node enlargement and de-novo CS-II patients). In this cohort, miRNA-371 level will be drawn at any timepoint after orchiectomy. Patients with initial CS-I and retroprertioneal relapse/ de-novo CS-II disease and normal miRNA-371 levels will undergo reassessment (repeat cross sectional imaging and miRNA level) after 6 weeks. If mass is stable and miRNA-371 level remains normal then patients will continue on surveillance. Patient will continue to be followed with miRNA levels with each conventional marker draw until 2 years, and followed according to standard of care guidelines until 5 years.
  Interventions: Other: Clinical Stage I with relapse, CSII Disease

INTERVENTIONS:
Other: Clinical Stage I Disease — Patients undergo blood sample collection during screening and throughout the study. Based on results, patients will undergo a primary RPLND surgery or standard surveillance. Surveillance will follow until year 5.
  Groups: Cohort 1
Other: Clinical Stage I with relapse, CSII Disease — Patients undergo blood sample collection during screening and throughout the study. Based on results, patients will undergo a primary RPLND surgery or reassessment and then surveillance will follow until year 5.
  Groups: Cohort 2

SUMMARY:
This study evaluates the accuracy of blood-based biomarker testing to predict the presence of active testicular cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To measure the accuracy of the blood-based biomarker miRNA-371 to predict pre-operatively the presence of active germ cell malignancy.

OUTLINE: This is an observational study.

Patients undergo blood sample collection during screening and throughout the study. Patients whose screening blood samples show elevated miRNA-371 proceed to standard RPLND surgery. Patients whose screening blood samples show normal levels of miRNA-371 undergo standard surveillance followed by standard RPLND surgery at the time of elevated miRNA-371 levels. Patients may also have their medical records reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Primary tumor excised by radical inguinal orchiectomy and pathology consistent with GCT (seminoma or NSGCT)
* Clinical stage of patient is either:

  * Stage I pure seminoma OR stage I pure seminoma with isolated retroperitoneal relapse or Stage IIA/B pure seminoma
  * Stage I NSGCT OR stage I NSGCT with isolated retroperitoneal relapse or Stage IIA/B NSGCT
* Suspected retroperitoneal disease: Lymphadenopathy in the retroperitoneum with no lymph node >3 cm in greatest dimension with no more than 2 nodes enlarged
* Axial abdominal/pelvic imaging (CT or MRI) and chest imaging (x-ray, CT or MRI) within 3 months of enrollment if stage I patient
* Axial abdominal/pelvic imaging (CT or MRI) and chest imaging (x-ray, CT or MRI) within 6 weeks of enrollment if stage II patient
* MiRNA-371 level drawn within 1 year after orchiectomy for stage I patients
* MiRNA-371 level drawn at any timepoint after orchiectomy for stage II patients
* Retroperitoneal lymphadenopathy must be within an RPLND template
* Biopsy of lymph node is not required, though if biopsy of the retroperitoneal node(s) was obtained, pathology must be consistent with GCT
* Serum Alpha Feto Protein (AFP), β-Human Chorionic Gonadotropin (HCG), Lactate Dehydrogenase (LDH) - per the local laboratory assay <1.5xlower normal level within 42 days (6 weeks) of enrollment
* Age ≥ 16 years
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Second primary malignancy
* History of receiving chemotherapy or radiotherapy
* Patients receiving any other investigational agent (s)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with testicular germ cell tumor
Sampling Method: Non-Probability Sample
Enrollment: 418 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2028-06-08 (Estimated); Study Completion 2028-12-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy of miRNA-371 to predict pre-operatively the presence of active germ cell malignancy | Through study completion, up to 5 years
  The positive predictive value of pre-operatively elevated miRNA-371 levels in predicting active GCT will be determined by pathologic review of RPLND specimens.

SECONDARY OUTCOMES:
The 2-year disease-free survival | Through study completion, up to 5 years
  Estimate the 2-year disease-free survival for patients who are miRNA negative at enrollment
Persistence of positive postoperative miRNA as a predictor of relapse at follow-up | Through study completion, up to 5 years
  Evaluate the relapse rate at follow-up in patients with positive postoperative miRNA after RPLND
Negative predictive value of negative pre-operative miRNA | Through study completion, up to 5 years
  Estimate the negative predictive value of negative pre-operative miRNA as confirmed by completing 2-year surveillance or pathological confirmation (i.e. biopsy or RPLND)

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Daneshmand, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California